CLINICAL TRIAL: NCT00753766
Title: Multifactorial Pre-Operative Intervention in Diabetes Mellitus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate participant recruitment
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-004-04F
Record Dates: First submitted 2008-09-12; First posted 2008-09-17 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus; Surgical Procedure, Unspecified
Keywords: A1c; Blood Glucose Management; Blood Pressure; Case Management; Diabetes Mellitus; Intervention study; Multifactorial; Peri-operative complications; Pre-operative
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multifactorial Intervention (Experimental): Mulitfactorial intervention - addressing glucose, blood pressure, lipids, smoking, nutrition and exercise.
  Interventions: Other: Multifactorial Intervention
- Usual care (No Intervention): Control group

INTERVENTIONS:
Other: Multifactorial Intervention
  Arms: Multifactorial Intervention

SUMMARY:
The purpose of this study is to advance the quality of care among inpatients with diabetes in the VHA. When patients with diabetes are admitted to the hospital, there is a greater chance that they will have a complication that lengthens their stay in the hospital. We are testing whether managing their diabetes before admission makes a difference in occurrence of in-hospital complications.

DETAILED DESCRIPTION:
Patients with diabetes that require hospitalization are at increased risk for morbidity and mortality, especially when undergoing surgery. There is some evidence that intensive glucose management during hospitalization may improve outcomes. However, no studies have evaluated intensive diabetes treatment before hospitalization.

Preliminary data from patients having vascular surgery show that those with diabetes have longer hospital stays, more frequent wound infections, and are more likely to require a return to the operating room when compared to patients without diabetes. In particular, insulin-treated patients have even greater peri-operative complications than non-insulin treated patients with diabetes. However, these data also suggest that a clinical trial to test the hypothesis that pre-operative intensive management has significant impact on peri-operative complications would require a very large number of participants to have adequate power.

Thus, our objective is to conduct a pilot and feasibility study to determine whether an intervention that involves intensive pre-operative diabetes management can be successfully implemented and to assess whether trends for benefit are observed. The results of this trial will support the conduct of a definitive study that tests the effectiveness of such an intervention in a larger sample of patients.

This is a randomized, parallel group clinical trial in insulin-treated patients with diabetes mellitus who have been scheduled for elective vascular surgery. We will randomize 46 participants diabetes mellitus: insulin-treated with HbA1c 7.5% or treated with oral agents with an elevated HbA1c who are scheduled for vascular surgery and in whom a 6 week pre-operative delay poses no substantial medical risks, as determined by the staff surgeon. We will exclude individuals with markedly elevated HbA1c or blood pressure; those with recently manifest cardiovascular disease, and those unable to attend regularly scheduled follow-up visits during the pre-operative period.

Participants will be randomized to either continue with usual care or participate in a multifactorial intervention conducted over a 6-week period. During the intervention period, participants will meet with a care manager and/or endocrinologist on at least 3 occasions and have telephone follow-up between these visits. They will receive instruction on lifestyle modifications; measure glucose and blood pressure at home (including the use of a continuous glucose monitoring device on 2 occasions), and receive care management to optimize glucose, blood pressure, and lipid lowering, as appropriate.

The primary outcome measure is the percent of screened participants that are eligible and choose participation Secondary end points will include: participant adherence with the study protocol, change from baseline in A1c and fructosamine, occurrence of wound infections in the 30-day peri-operative period, a composite of death from cardiovascular causes, non-fatal myocardial infarction, coronary artery bypass grafting, percutaneous coronary intervention, nonfatal stroke, or amputation as a result of peripheral ischemia; length of hospital stay; and rate of return to the operating room.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus
* A1c 7.5%,
* Scheduled elective vascular surgery that may be safely deferred for 6 weeks
* Surgeon's approval to participate

Exclusion Criteria:

* Hemoglobin A1c >14% (This criterion was included since, once identified, such a patient warrants improved glucose control and can not be ethically entered into a trial where there is a 50% chance of being assigned to usual care)
* Myocardial infarction in prior 6 months
* Cerebrovascular disease in prior 6 months
* Active cancer requiring ongoing treatment
* Severe psychiatric disease limiting ability to comply with protocol
* Unable to attend follow up appointments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul R. Conlin, MD, Principal Investigator — VA Boston Healthcare System West Roxbury Campus, West Roxbury, MA

RESULTS

PARTICIPANT FLOW:
Groups:
- Multifactorial Intervention: Mulitfactorial intervention - included addressing glucose, blood pressure, lipids, smoking, nutrition and exercise.
Period: Overall Study
Arm/Group | Multifactorial Intervention | Usual Care
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: The one participant who entered the trial was assigned to the Multifactorial Intervention group but was withdrawn from the study for safety reasons, and their data could not be analyzed. There were -0- participants enrolled in the Usual Care group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Multifactorial Intervention | Usual Care | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent of Screened Participants That Are Eligible and Choose Participation
Time Frame: 6 weeks
Population: The one participant who entered the trial was assigned to the Multifactorial Intervention group but was withdrawn from the study for safety reasons, and very limited data could be analyzed. There were -0- participants enrolled in the Usual Care group.
Measure: Number; unit: percentage of potential participants
Arm/Group | Multifactorial Intervention | Usual Care
Number analyzed (Participants) | 1 | 0
percentage of potential participants | 100 |

2. Secondary Outcome: Percentage of Participants With Full Adherence to the Study Protocol (i.e. Attending Study Visits, CGMS Studies)
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Number; unit: percent of participants
Groups:
- Multifactorial Intervention: Mulitfactorial intervention - addressing glucose, blood pressure, lipids, smoking, nutrition and exercise.
  Multifactorial Intervention
Arm/Group | Multifactorial Intervention | Usual Care
Number analyzed (Participants) | 1 | 0
percent of participants | 0 |

3. Secondary Outcome: Percentage of Participants Not Completing the Protocol Due to the Need for Urgent Surgery and/or Treatment-related Complications
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Number; unit: percent of participants
Arm/Group | Multifactorial Intervention | Usual Care
Number analyzed (Participants) | 1 | 0
percent of participants | 100 |

4. Secondary Outcome: Change in A1c From Baseline to Pre-admission (A1c is the Standard Parameter to Assess Chronic Glucose Control])
Description: A1c measured at two time points - baseline and 6 weeks later (pre-admission). This parameter is the difference between those two time points.
Time Frame: 6 weeks
Population: The one participant who entered the trial was assigned to the Multifactorial Intervention group but was withdrawn from the study for safety reasons, and data for this parameter were not collected. There were -0- participants enrolled in the Usual Care group.
Arm/Group | Multifactorial Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Occurrence of Wound Infection in the 30 Day Post-operative Period
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Multifactorial Intervention | Usual Care
Number analyzed (Participants) | 1 | 0
Participants | 0 |

6. Secondary Outcome: Length of Hospital Stay
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Number; unit: days
Arm/Group | Multifactorial Intervention | Usual Care
Number analyzed (Participants) | 1 | 0
days | 6 |

7. Secondary Outcome: Number of Participants Who Experience a Composite of Death From Cardiovascular Cause, Non-fatal Myocardial Infarction, Coronary Artery Bypass Grafting, Percutaneous Coronary Intervention, Nonfatal Stroke, or Amputation as a Result of Peripheral Ischemia
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Multifactorial Intervention | Usual Care
Number analyzed (Participants) | 1 | 0
Participants | 0 |

8. Secondary Outcome: Percentage of Participants Who Need to Return to the Operating Room
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Number; unit: percent of participants
Arm/Group | Multifactorial Intervention | Usual Care
Number analyzed (Participants) | 1 | 0
percent of participants | 0 |

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: The one participant who entered the trial was assigned to the Multifactorial Intervention group but was withdrawn from the study for safety reasons, and very limited data could be analyzed. There were -0- participants enrolled in the Usual Care group.
Arm/Group | Multifactorial Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No